CLINICAL TRIAL: NCT06341816
Title: Regulation of Treatment According to Venous Load Ultrasound Score (VEXUS) in Patients Followed in Intensive Care Due to Heart Failure
Brief Title: Treatment According to Venous Excess Ultrasound Score in Patients With Heart Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ayse Belin Ozer, Prof. Dr., Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VEXUS2
Record Dates: First submitted 2024-03-20; First posted 2024-04-02 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure; Acute Kidney Injury
MeSH Terms: conditions — Heart Failure; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): In the conventional group, heart failure treatment will be managed according to classical physical examination (e.g. peripheral edema, rales) and laboratory methods (pro-BNP). e.g. fluid restriction, diuretic therapy, etc.
  Interventions: Other: VEXUS score; Diagnostic Test: NGAL
- VEXUS (Active Comparator): In the vexus group, heart failure treatment will be given in a way that will reduce the vexus score. e.g. fluid restriction, diuretic therapy, etc.
  Interventions: Other: VEXUS score; Diagnostic Test: NGAL

INTERVENTIONS:
Other: VEXUS score — The VExUS score is obtained as follows: VEXUS 0: IVC < 20mm; VEXUS 1: IVC ≥ 20mm with normal patterns or mild abnormalities; VEXUS 2: IVC ≥ 20mm with severe abnormality in at least one pattern and VEXUS 3: IVC ≥ 20mm and severe abnormalities in multiple patterns.
Diagnostic Test: NGAL — Neutrophil gelatinase-associated lipocalin

SUMMARY:
Heart failure is a syndrome that progresses with symptoms and signs caused by cardiac dysfunction and results in a shortened life expectancy (1). Acute heart failure resulting in hospitalization is a significant cause of morbidity and mortality. With the increase in the severity of the disease and rapid advances in the treatment of heart failure, these patients are frequently hospitalized and monitored in intensive care. (2) Five years after diagnosis, mortality can be up to 67%. Additionally, it is known that patients with heart failure are hospitalized on average once a year after diagnosis. (3) In a multicenter study, it constituted 14% of 3000 cardiac patients admitted to intensive care units. Additionally, due to longer ICU stays, these patients accounted for 33% of total inpatient days. An increasing number of heart failure patients require intensive care due to respiratory failure, regardless of left ventricular ejection fraction. Heart failure accounts for approximately one-third of patient days in intensive care units, and this burden is increasing. This shows that attention should be paid to the quality of care for patients requiring critical care. (2) Multidisciplinary programs have been implemented to deal with the high prevalence. However, the optimal follow-up frequency is unknown. Therefore, some tools are needed to improve patient prognosis (3).

Neutrophil gelatinase-associated lipocalin (NGAL) is a biomarker whose values in both urine and plasma have been associated with acute kidney injury (AKI). Although NGAL is an early specific biomarker for AKI, it has not yet come into routine use, but is frequently used in clinical and experimental studies (4).

Venous load ultrasonography score (VExUS) is a new systemic congestion scoring method based on inferior vena cava dilation and pulsed wave Doppler (PW-Doppler) morphology of the hepatic, portal and renal veins. It has been proposed as a score to assess systemic congestion.

DETAILED DESCRIPTION:
Patients will be randomized according to the sealed envelope method. While classical heart failure fluid management will be applied to patients in the conventional group, diuretic treatment will be given to the vexus group in a way that will reduce the vexus score, and the drugs and doses used in this treatment will be recorded.

The development of acute renal failure in patients will be determined according to KDIGO criteria, but confirmation will be made with NGAL.

Patients will be divided into two groups: those treated according to the VEXUS score and those treated simultaneously with VEXUS by a second experienced person (INTENSIVE CARE SPECIALIST) but treated conservatively. Patients' vital parameters, complete blood count, biochemistry, coagulation, arterial blood gas, procalcitonin, CRP, troponin, pro-BNP levels on Day 1 and Day 5 will be noted, and distensibility will be detected by USG on Days 1 and 5 among those with an IVC diameter < 2 cm. or collapsibility index, and for those > 2cm, VEXUS score will be calculated. In addition, EF, TAPSE, presence of pleural effusion or B-Line, renal resistive index, renal pulsatility index will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a life expectancy of more than 24 hours
* >18 age

Exclusion Criteria:

* Poor abdominal echogenicity
* age < 18
* postoperative patients,
* intoxications,
* life expectancy is less than 24 hours,
* pregnancy,
* intraperitoneal pressure > 15 mm Hg,
* obstructive renal failure or suspected,
* presence of renal artery stenosis,
* patients who have had liver and kidney transplants,
* Presence of liver and kidney tumors,
* patients receiving dialysis treatment,
* single kidney and other kidney abnormalities,
* presence of acute mesenteric ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-25 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
acute kidney injury | first week
  it will evaluate according to KDİGO criteria
mortality | in 28 days
  in 28 days mortality

IPD SHARING:
Plan to Share IPD: No